CLINICAL TRIAL: NCT00226928
Title: Psychosocial Treatment Effects on Cancer Survival
Brief Title: Psychosocial Treatment for Improving Chances of Survival in Women With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, David Spiegel, Jack, Lulu & Sam Willson Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R01MH047226 (NIH); R01MH047226 (NIH); DAHBR HB-C
Record Dates: First submitted 2005-09-12; First posted 2005-09-27 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: Stage IIIB, IV, Recurrent, and Metastatic Breast Cancer
MeSH Terms: conditions — Recurrence; Breast Neoplasms | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Supportive-Expressive Group Therapy plus education
Behavioral: Education

SUMMARY:
This study will investigate the influence of psychosocial treatment on psychological outcomes and survival among women with metastatic or recurrent breast cancer.

DETAILED DESCRIPTION:
The objective of this study is to investigate the influence of psychosocial treatment on psychological outcomes and survival among women with metastatic/recurrent breast cancer.

ELIGIBILITY:
Inclusion Criteria:

Women were eligible for the study if they had documented metastatic or recurrent breast cancer, were proficient enough in English to be able to complete questionnaires and participate in a support group, were living in the Greater San Francisco Bay Area, and had a Karnofsky score of at least 70%.19 Exclusion Criteria:

Women were excluded if they had any of the following risk factors: positive supraclavicular lymph nodes as the only metastatic lesion at the time of initial diagnosis; active non-breast cancers within the past 10 years; or other concurrent medical conditions likely to influence short-term survival. Basal cell or squamous cell carcinomas of the skin, in situ cancer of the cervix, or melanoma with a Breslow depth less than 0.76 mm were allowed.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Study Completion 2005-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Spiegel, M.D., Principal Investigator — Stanford University

REFERENCES:
- [Result] Butler LD, Field NP, Busch AL, Seplaki JE, Hastings TA, Spiegel D. Anticipating loss and other temporal stressors predict traumatic stress symptoms among partners of metastatic/recurrent breast cancer patients. Psychooncology. 2005 Jun;14(6):492-502. doi: 10.1002/pon.865. PMID 15452896
- [Result] Giese-Davis J, Sephton SE, Abercrombie HC, Duran RE, Spiegel D. Repression and high anxiety are associated with aberrant diurnal cortisol rhythms in women with metastatic breast cancer. Health Psychol. 2004 Nov;23(6):645-50. doi: 10.1037/0278-6133.23.6.645. PMID 15546233
- [Result] Turner-Cobb JM, Koopman C, Rabinowitz JD, Terr AI, Sephton SE, Spiegel D. The interaction of social network size and stressful life events predict delayed-type hypersensitivity among women with metastatic breast cancer. Int J Psychophysiol. 2004 Nov;54(3):241-9. doi: 10.1016/j.ijpsycho.2004.05.010. PMID 15331215
- [Result] Blake-Mortimer JS, Sephton SE, Carlson RW, Stites D, Spiegel D. Cytotoxic T lymphocyte count and survival time in women with metastatic breast cancer. Breast J. 2004 May-Jun;10(3):195-9. doi: 10.1111/j.1075-122X.2004.21290.x. PMID 15125744
- [Result] Butler LD, Koopman C, Cordova MJ, Garlan RW, DiMiceli S, Spiegel D. Psychological distress and pain significantly increase before death in metastatic breast cancer patients. Psychosom Med. 2003 May-Jun;65(3):416-26. doi: 10.1097/01.psy.0000041472.77692.c6. PMID 12764215
- [Result] Koopman C, Nouriani B, Erickson V, Anupindi R, Butler LD, Bachmann MH, Sephton SE, Spiegel D. Sleep disturbances in women with metastatic breast cancer. Breast J. 2002 Nov-Dec;8(6):362-70. doi: 10.1046/j.1524-4741.2002.08606.x. PMID 12390359
- [Result] Giese-Davis J, Koopman C, Butler LD, Classen C, Cordova M, Fobair P, Benson J, Kraemer HC, Spiegel D. Change in emotion-regulation strategy for women with metastatic breast cancer following supportive-expressive group therapy. J Consult Clin Psychol. 2002 Aug;70(4):916-25. doi: 10.1037//0022-006x.70.4.916. PMID 12182275
- [Result] Sephton SE, Koopman C, Schaal M, Thoresen C, Spiegel D. Spiritual expression and immune status in women with metastatic breast cancer: an exploratory study. Breast J. 2001 Sep-Oct;7(5):345-53. doi: 10.1046/j.1524-4741.2001.20014.x. PMID 11906445
- [Result] Classen C, Butler LD, Koopman C, Miller E, DiMiceli S, Giese-Davis J, Fobair P, Carlson RW, Kraemer HC, Spiegel D. Supportive-expressive group therapy and distress in patients with metastatic breast cancer: a randomized clinical intervention trial. Arch Gen Psychiatry. 2001 May;58(5):494-501. doi: 10.1001/archpsyc.58.5.494. PMID 11343530
- [Result] Turner-Cobb JM, Sephton SE, Koopman C, Blake-Mortimer J, Spiegel D. Social support and salivary cortisol in women with metastatic breast cancer. Psychosom Med. 2000 May-Jun;62(3):337-45. doi: 10.1097/00006842-200005000-00007. PMID 10845347
- [Result] Butler LD, Koopman C, Classen C, Spiegel D. Traumatic stress, life events, and emotional support in women with metastatic breast cancer: cancer-related traumatic stress symptoms associated with past and current stressors. Health Psychol. 1999 Nov;18(6):555-60. doi: 10.1037//0278-6133.18.6.555. PMID 10619528
- [Result] Koopman C, Hermanson K, Diamond S, Angell K, Spiegel D. Social support, life stress, pain and emotional adjustment to advanced breast cancer. Psychooncology. 1998 Mar-Apr;7(2):101-11. doi: 10.1002/(SICI)1099-1611(199803/04)7:23.0.CO;2-3. PMID 9589508
- [Result] Classen C, Koopman C, Angell K, Spiegel D. Coping styles associated with psychological adjustment to advanced breast cancer. Health Psychol. 1996 Nov;15(6):434-7. doi: 10.1037//0278-6133.15.6.434. PMID 8973923
- [Result] Sephton SE, Sapolsky RM, Kraemer HC, Spiegel D. Diurnal cortisol rhythm as a predictor of breast cancer survival. J Natl Cancer Inst. 2000 Jun 21;92(12):994-1000. doi: 10.1093/jnci/92.12.994. PMID 10861311
- [Derived] Butler LD, Koopman C, Neri E, Giese-Davis J, Palesh O, Thorne-Yocam KA, Dimiceli S, Chen XH, Fobair P, Kraemer HC, Spiegel D. Effects of supportive-expressive group therapy on pain in women with metastatic breast cancer. Health Psychol. 2009 Sep;28(5):579-87. doi: 10.1037/a0016124. PMID 19751084
- [Derived] Spiegel D, Butler LD, Giese-Davis J, Koopman C, Miller E, DiMiceli S, Classen CC, Fobair P, Carlson RW, Kraemer HC. Effects of supportive-expressive group therapy on survival of patients with metastatic breast cancer: a randomized prospective trial. Cancer. 2007 Sep 1;110(5):1130-8. doi: 10.1002/cncr.22890. PMID 17647221